CLINICAL TRIAL: NCT02220868
Title: Sofosbuvir, Ribavirin, for the Treatment of Chronic Hepatitis C Virus Genotype 1 in HIV-Coinfected Patients Receiving Fixed Dose Co-formulation Emtricitabine/ Tenofovir/Cobicistat/Elvitegravir: A Pilot Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Saint Michael's Medical Center (Other)
Responsible Party: Principal Investigator, Jihad Slim, MD, Chief and Prgram Director, Infectious Diseases, Saint Michael's Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IN-US-334-1527
Record Dates: First submitted 2014-08-18; First posted 2014-08-20 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2015-11

CONDITIONS: Hepatitis C Infection; HIV Infection
Keywords: HIV; HCV; DAA
MeSH Terms: conditions — Hepatitis C; HIV Infections | interventions — Sofosbuvir; Ribavirin; Elvitegravir, Cobicistat, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sofossbuvir, Riabvirin, Stribild (Other): Open-Label SIngle Arm of Sofosbuvir, Ribavirin and Stribild
  Interventions: Drug: Sofosbuvir, Ribavirin, and Stribild

INTERVENTIONS:
Drug: Sofosbuvir, Ribavirin, and Stribild

SUMMARY:
The protocol will study the safety and efficacy of using sofosbuvir and ribavirin for the treatment of hepatitis c in patients taking stribild.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the safety, efficacy and pharmacokinetics of sofosbuvir 400mg once daily plus ribavirin 1000-1200 mg daily in HIV-infected patients on fixed dose co-formulation emtricitabine/tenofovir/cobicistat/elvitegravir (Stribild).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Chronic HCV genotype 1 infection
* Receiving emtricitabine/tenofovir/cobicistat/elvitegravir for at least 8 weeks.
* CD4 count >200 cells/mm3 at screening and no CD4 count <200 in previous 12 weeks
* HIV RNA PCR <50 copies/ml at screening and no HIV RNA PCR > 200 copies/ml in previous 12 weeks

Exclusion Criteria:

* History of integrase inhibitor resistance
* History of integrase inhibitor failure
* Absolute neutrophil counts under 1500/mm3 ( Black/ African Americans <1200/mm3
* Patients with cirrhosis
* Platelet count under 90,000 per cubic millimeter
* Hemoglobin levels <11 gm/dl in women or <12 gm/dl in men
* Previous treatment with a DAA
* Hepatocellular carcinoma
* AFP>100 ng/mL
* hepatitis B virus (HBsAg positive)
* Evidence of decompensated liver disease including, but not limited to, a history of presence of clinical ascites, bleeding varices, or hepatic encephalopathy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-07; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
• SVR,12 defined as undetectable HCV RNA levels for 12 weeks after the completion of therapy | 12 weeks post treatment
  patients who have achieved non-detectable HCV levels 12 weeks post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jihad Slim, MD, Principal Investigator — Saint Michael's Medical Center
Locations (1):
- Saint Michael's Medical Center, Newark, New Jersey, United States